CLINICAL TRIAL: NCT04541784
Title: Effectiveness of a Multidimensional Mobile App Intervention "WOMAN-PRO III" to Reduce Postsurgical Symptom Induced Distress in Patients With Vulvar Neoplasia: A Mixed Methods Project
Brief Title: Effectiveness of an App Intervention to Reduce Postsurgical Symptom Distress in Patients With Vulvar Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St.Gallen University of Applied Sciences (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); Cantonal Hospital of Lucerne (Unknown); Regional Hospital of Lugano (Unknown); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Andrea Kobleder, Principal Investigator, St.Gallen University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WOMAN-PRO III
Record Dates: First submitted 2020-08-12; First posted 2020-09-09 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Vulvar Neoplasm
Keywords: mHealth; Postsurgical symptoms; Distress; Uncertainty; Mixed methods
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers and the statistician will be blinded to treatment assignment to prevent ascertainment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 counselling sessions with gynaecology-oncology nurses (Active Comparator): Patients randomized to the control group will receive standardized care, 3 counselling sessions with a gynaecology-oncology nurse and written information at three points in time during 6 months after diagnosis/surgery.
  Interventions: Other: Three counselling sessions with gynaecology-oncology nurses
- Mobile app and 3 counselling sessions (WOMAN-PROIII) (Experimental): Standardized care and three counselling sessions with a gynaecology-oncology nurse and the use of the mobile app "WOMAN-PRO III". Counselling sessions will take place at 3 points in time during 6 months after diagnosis/surgery. Additionally, the gynaecology-oncology nurse will instruct the patient to use the mobile app. It includes a diary for symptom assessment and gives graphical feedback. Further, the app includes disease and treatment related information. If a symptom occurs the app will give an evidence-based recommendation (Kobleder et al., 2016). The patients can use the app whenever they want for a period of six months.
  Interventions: Other: WOMAN-PRO III

INTERVENTIONS:
Other: WOMAN-PRO III — Standardized care and three counselling sessions with a gynaecology-oncology nurse and the use of the mobile app "WOMAN-PRO III".
  Arms: Mobile app and 3 counselling sessions (WOMAN-PROIII)
Other: Three counselling sessions with gynaecology-oncology nurses — Standardized care, three counselling sessions with a gynaecology-oncology nurse.
  Arms: 3 counselling sessions with gynaecology-oncology nurses

SUMMARY:
Despite great advances in surgical therapy in the last decades, symptom relief for women with vulvar neoplasia (vulvar cancer and pre-stage of vulvar cancer) is still not optimal. Guidelines of the National Comprehensive Cancer Network recommend using electronic communication media, e.g. applications ("apps") to relieve symptom distress and foster self-management. However, little is known on how effective these communication technologies are, especially in the field of a rare cancer disease like vulvar neoplasia. This mixed methods project aims to examine the effectiveness of a multidimensional mobile app intervention ("WOMAN-PRO III") focusing on possible improvements due to the new mobile app intervention, which consists of three counselling sessions with a gynaecologic-oncology nurse and the use of the mobile app whenever women want for a period of six months, the online version of the "WOMAN-PRO" diary for symptom assessment, the opportunity to send the data to the gynaecology-oncology nurse, disease and treatment related information and evidence-based recommendations, relevant contact data and a chat function for the anonymous exchange with peers (intervention group) compared to three counselling sessions with a gynaecologic-oncology nurse, where they receive written information (control group). Effectiveness will be examined with respect to symptom induced distress, uncertainty and cost effectiveness in women with vulvar neoplasia after surgical treatment across time.

The objective of the qualitative study is to assess women's perceived uncertainty and the acceptability, usability, strengths and weaknesses of the mobile app intervention ("WOMAN-PRO III") from patients' and gynaecology-oncology nurses' perspective.

DETAILED DESCRIPTION:
Vulvar neoplasia - incidence, symptoms and disease's management Although being a rare cancer disease, the incidence of vulvar neoplasia is increasing with a current incidence rate of 3.6 / 100.000 for women with vulvar cancer (Buttmann-Schweiger et al., 2015) and 7 / 100.000 for women with VIN (Anders, Riethdorf, & Löning, 2001). Due to the disease itself and treatment side effects women suffer from a high number of postsurgical symptoms and related distress, such as pain, swelling, or uncertainty (Jefferies & Clifford, 2012; Philp, Mellon, Barnett, D'Abrew, & White, 2017; Senn et al., 2011). Results from literature suggest that women have unmet support needs as talking to healthcare professionals is perceived as difficult and information given by healthcare professionals is described as conflicting and inadequate (Philp et al., 2017). The high symptom prevalence and related distress reported uncertainty as well as the perceived lack of supportive care can lead to hospital readmissions and consequently to the generation of high healthcare costs.

To overcome this lack of supportive care, guidelines focusing on vulvar neoplasia recommend an integrative approach including skilled nursing as a key factor for patient management (Royal College of Obstetricians and Gynaecologists, 2014). Specialist nurses, i.e. Advanced Practice Nurses (APN) can, therefore, play an important role in caring for women with vulvar neoplasia, as shown in the study of Raphaelis et al. (2018) where women received written information and counselling sessions from APNs. However, gaps remain especially in women's disease management beyond the walls of the clinic. Therefore, supportive care interventions are requested to promote women's self-management, especially at home. One possibility might be the use of e-health.

E-health - the changing nature of self-help: E-health has come to be an important avenue for supporting self-management. One integral part of the subject area of e-health is m-health. Within the healthcare system the aim of m-health is to provide electronic solutions on mobile devices, which is also described in the WHO definition of m-health: "M-health covers medical and public health practice supported by mobile devices, such as mobile phones, patient monitoring devices, personal digital assistants (PDAs), and other wireless devices" (World Health Organization, 2011). It is expected to contribute to patients' empowerment as they could take a more active role (European Commission, without date). Especially in chronic disease management, m-health interventions could play an important role in providing information and enabling communication without spatial and temporal restrictions.

Significance: This research will contribute significantly to the knowledge about effects of mobile app interventions in gynaecologic oncology, especially with regard to a reduction of symptom induced distress and improvement of uncertainty in a stigmatized disease like vulvar neoplasia.

Objectives: Primary Objective The study seeks primarily to examine the effectiveness of a multidimensional mobile app intervention, which consists of the use of the mobile app whenever women want for a period of six months and three counselling sessions with a gynaecology-oncology nurse ("WOMAN-PRO III") on symptom induced distress, uncertainty and cost-effectiveness in women with vulvar neoplasia after surgical treatment across time compared to three counselling sessions with a gynaecology-oncology nurse and written information. The secondary objective is to explore women's perceived uncertainty as well as the mobile app's acceptability, usability, strengths and weaknesses by assessing participants' and gynaecology-oncology nurses' experiences.

Methods: We use an explanatory-sequential design (Creswell & Plano Clark, 2017) to examine the effectiveness of the mobile-app intervention ("WOMAN-PRO III"). Thus, quantitative findings can be explained by means of qualitative results (Creswell & Plano Clark, 2017). Therefore, Phase 1 of this project will consist of a randomized controlled trial (RCT) with an intervention and control arm. Phase 2 is a subsequent qualitative study aiming to explore (1) women's meaning of uncertainty and (2) the mobile app intervention's ("WOMAN PRO III") acceptability, usability, strengths and weaknesses from patients' and gynaecology-oncology nurses' perspective.

Sample and setting: 100 Patients, with an estimated rate of 20% loss to follow-up and drop-out will be recruited continuously in four Swiss hospitals (Bern, Lucerne, Lugano, St.Gallen) to have in the end a total sample of 80 patients for analysis.

Recruitment: From May 1st, 2019 until January31st, 2021 patients will be consecutively invited by a gynaecologist or a nurse to participate in the study after initial diagnosis at the hospital.

Data collection: Will be conducted in the control group via paper-based questionnaires and in the intervention group via paper-based questionnaires and additionally via app. Patients will be asked to complete questionnaires at three points in time:

* Diagnosis / before surgical intervention (t0),
* day seven after surgery (t1),
* and month six after surgery (t2). Sample size: Statistical significance is defined as α = 0.05, power is defined as 80%. Assuming a 20% rate of loss to follow-up and drop-out, with a sampling ratio of 1 a total of 100 female patients with surgically treated VIN/VC will be necessary to start the randomized control trial to gain a total sample of 80 patients for analysis.

Planned analyses: Patients will be analyzed within their assigned groups (intention to treat) based on frequencies and descriptive statistics. Changes in symptom induced distress (frequency of symptoms, items and subscores) will be analyzed using mixed linear regression analysis, taking into account the longitudinal nature of the data (t0, t1, t2), and data clustering within centers. Fixed variables will be study group, point of time, and their interaction. The variables 'patient', nested under the respective 'center', will be entered as a random effect. To find out time-specific differences between the patient groups post-hoc tests will be performed. Uncertainty, our secondary outcome, will be analyzed similarly. Statistical analysis will be provided by a professional statistician, using IBM SPSS Version 24.

Qualitative study: After 6 months of collecting data for the RCT, a qualitative study will be started aiming to explore (1) women's perceived meaning and interaction concerning uncertainty and (2) the mobile app intervention's ("WOMAN PRO III") acceptability, usability, strengths and weaknesses from patients' and gynaecology-oncology nurses' perspective. Therefore, interviews will be conducted with women participating in the RCT and women who agreed to only participate in the qualitative study. Further, a focus group will be conducted with gynaecology-oncology nurses involved in the intervention tested.

Sample and setting: Women who have participated in Phase one of the mixed methods study will be considered as suitable to give insights about their meaning of uncertainty. As well, women who were not interested in participating in the RCT, but declared interest in participating in the qualitative study, are found to be eligible. Participants of the intervention and gynaecology-oncology nurses involved in the mobile app intervention (6 - 8 nurses) are considered eligible to deliver information about the mobile app intervention's ("WOMAN PRO III") acceptability, usability, strengths and weaknesses. It can be assumed, that with interviewing about 15 patients and involving 6 - 8 gynaecology-oncology nurses a first data saturation can be achieved.

Recruitment: Six months after surgery (t2) patients will be asked by a nurse not involved in the patients' treatment to indicate their willingness to participate in an individual interview. All gynaecology-oncology nurses involved in the mobile app intervention will be asked to participate in the focus group interview.

Data collection: The patient interviews and the focus group with the gynaecology-oncology nurses will be conducted by using interview guides consisting of open-ended questions. The interviews and the focus group will last about an hour. Patients' interviews will take place at the participant's home or in the clinical setting according to patient's preferences. The focus group interview will be held at a research institute. ¨ Data analysis: Data of the patient interviews and the focus group will be recorded, anonymized and transcribed verbatim (Dresing & Pehl, 2011) and analyzed using open, axial and selective coding as proposed by Corbin & Strauss (2015). The data analysis process will be conducted by researchers with extended experience in qualitative research and assisted by MAXQDA 2018 (VERBI GmbH, Berlin).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis VIN or vulvar cancer (primary diagnosis or recurrent neoplasia)
* Surgical treatment of VIN or vulvar cancer in one of the designated hospitals
* Sufficient knowledge of the German/Italian language (writing and speaking at level B1)
* Having a smartphone (e.g. iPhone, Samsung), tablet (e.g. iPad) or laptop (e.g. MacBook) for women participating in the quantitative study
* Informed Consent as documented by signature (Appendix Informed Consent Form)

Exclusion Criteria:

* Patients being judged by a physician or by a gynaecology-oncology nurse specialist as not being capable to participate in the trial and to complete the questionnaire due to:
* Cognitive, linguistic, emotional or physical reasons
* A present psychiatric treatment by reason of a main psychiatric diagnosis and the intake of psychopharmacological drugs
* Terminal illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change of symptom induced distress | Between diagnosis / before surgical treatment (t0), day seven post-surgery (t1) and month six post-surgery (t2)
  Measured with the "WOMAN-PRO" symptom diary. This instrument focuses on patients' post-surgical symptom experience, regarding frequency and distress. The instrument consists of 36 items covering four domains. On average a patient needs 20 minutes to complete the diary. The instrument showed an excellent item validity (Cronbach's alpha ranging between 0.74 and 0.90) and scale content validity (CVI=1.0) (Senn et al., 2013).

SECONDARY OUTCOMES:
Uncertainty | Between diagnosis / before surgical treatment (t0), day seven post-surgery (t1) and month six post-surgery (t2)
  Measured with the Mishel Uncertainty in Illness Scale (MUIS). The MUIS is a 30-item scale assessing uncertainty in symptomatology, diagnosis, treatment, relationship with care-givers and planning for the future for patients with cancer. Internal consistency showed a multi-attributed ambiguity alpha ranging from 0.89-0.91 and an unpredictability alpha from 0.64-0.72. Scale development based on theoretical framework of cognitive appraisal model and perceived uncertainty in illness model as well as interviews with patients and health provider review. Factors were identified by factor analysis and confirmed by replication out of sample (Mishel, 1981).
Cost effectiveness | During a period of 6 months after diagnosis/surgery
  Measured by means of a within-trial analysis, comparing direct costs and six-month outcomes of patients randomized to the intervention versus control group. The economic evaluation will consist of a cost-effectiveness analysis (CEA) which includes treatment expenses (intervention costs) and the identified differences in symptom distress.

OTHER OUTCOMES:
Sociodemographic data | At diagnosis/before surgery (t0)
  Collected using an 11-item paper-based questionnaire. Items will include age, marital status, number of children, education, employment status, living situation, post-surgical wound management at home and health insurance.
Medical data | At diagnosis/before surgery (t0)
  Collected by the gynaecology-oncology nurse using a 16-item paper- based questionnaire concerning diagnosis, cancer stage, initial and wound treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Switzerland (4):
  - Cantonal Hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Regional Hospital of Lugano, Lugano, Canton Ticino
  - University Hospital of Bern, Bern
  - Cantonal Hospital of Lucerne, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broglia E, Millings A, Barkham M. Comparing counselling alone versus counselling supplemented with guided use of a well-being app for university students experiencing anxiety or depression (CASELOAD): protocol for a feasibility trial. Pilot Feasibility Stud. 2017 Jan 23;3:3. doi: 10.1186/s40814-016-0119-2. eCollection 2017. PMID 28127442
- [Background] Buttmann-Schweiger N, Klug SJ, Luyten A, Holleczek B, Heitz F, du Bois A, Kraywinkel K. Incidence patterns and temporal trends of invasive nonmelanotic vulvar tumors in Germany 1999-2011. A population-based cancer registry analysis. PLoS One. 2015 May 28;10(5):e0128073. doi: 10.1371/journal.pone.0128073. eCollection 2015. PMID 26020540
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] U.S. Department of Health and Human Services FDA Center for Drug Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Biologics Evaluation and Research; U.S. Department of Health and Human Services FDA Center for Devices and Radiological Health. Guidance for industry: patient-reported outcome measures: use in medical product development to support labeling claims: draft guidance. Health Qual Life Outcomes. 2006 Oct 11;4:79. doi: 10.1186/1477-7525-4-79. PMID 17034633
- [Background] Gray HJ. Advances in vulvar and vaginal cancer treatment. Gynecol Oncol. 2010 Jul;118(1):3-5. doi: 10.1016/j.ygyno.2010.04.011. Epub 2010 May 15. No abstract available. PMID 20471671
- [Background] Graziottin A, Serafini A. HPV infection in women: psychosexual impact of genital warts and intraepithelial lesions. J Sex Med. 2009 Mar;6(3):633-45. doi: 10.1111/j.1743-6109.2008.01151.x. Epub 2009 Jan 13. PMID 19170869
- [Background] Jefferies H, Clifford C. Invisibility: the lived experience of women with cancer of the vulva. Cancer Nurs. 2012 Sep-Oct;35(5):382-9. doi: 10.1097/NCC.0b013e31823335a1. PMID 22067693
- [Background] Kaushik S, Pepas L, Nordin A, Bryant A, Dickinson HO. Surgical interventions for high-grade vulval intraepithelial neoplasia. Cochrane Database Syst Rev. 2014 Mar 4;2014(3):CD007928. doi: 10.1002/14651858.CD007928.pub3. PMID 24596022
- [Background] Kobleder A, Raphaelis S, Glaus A, Fliedner M, Mueller MD, Gafner D, Gehrig L, Senn B. Recommendations for symptom management in women with vulvar neoplasms after surgical treatment: An evidence-based guideline. Eur J Oncol Nurs. 2016 Dec;25:68-76. doi: 10.1016/j.ejon.2016.10.003. Epub 2016 Oct 22. PMID 27865255
- [Background] Leermakers ME, Pleunis N, Boll D, Hermans RH, Ezendam NP, Pijnenborg JM. High Incidence of Erysipelas After Surgical Treatment for Vulvar Carcinoma: An Observational Study. Int J Gynecol Cancer. 2016 Mar;26(3):582-7. doi: 10.1097/IGC.0000000000000625. PMID 26807636
- [Background] McFadden KM, Sharp L, Cruickshank ME. The prospective management of women with newly diagnosed vulval intraepithelial neoplasia: clinical outcome and quality of life. J Obstet Gynaecol. 2009 Nov;29(8):749-53. doi: 10.3109/01443610903191285. PMID 19821671
- [Background] Mishel MH. The measurement of uncertainty in illness. Nurs Res. 1981 Sep-Oct;30(5):258-63. PMID 6912987
- [Background] Philp S, Mellon A, Barnett C, D'Abrew N, White K. The road less travelled: Australian women's experiences with vulval cancer. Eur J Cancer Care (Engl). 2017 Jan;26(1). doi: 10.1111/ecc.12465. Epub 2016 Feb 18. PMID 26892880
- [Background] Raphaelis S, Mayer H, Ott S, Mueller MD, Steiner E, Joura E, Senn B. The impact of written information and counseling (WOMAN-PRO II Program) on symptom outcomes in women with vulvar neoplasia: A multicenter randomized controlled phase II study. Gynecol Oncol. 2017 Jul;146(1):114-122. doi: 10.1016/j.ygyno.2017.04.024. Epub 2017 May 5. PMID 28483270
- [Background] Raphaelis S, Mayer H, Ott S, Hornung R, Senn B. Effects of Written Information and Counseling on Illness-Related Uncertainty in Women With Vulvar Neoplasia. Oncol Nurs Forum. 2018 Nov 1;45(6):748-760. doi: 10.1188/18.ONF.748-760. PMID 30339152
- [Background] Senn B, Gafner D, Happ MB, Eicher M, Mueller MD, Engberg S, Spirig R. The unspoken disease: symptom experience in women with vulval neoplasia and surgical treatment: a qualitative study. Eur J Cancer Care (Engl). 2011 Nov;20(6):747-58. doi: 10.1111/j.1365-2354.2011.01267.x. Epub 2011 Jul 19. PMID 21771133
- [Background] Senn B, Eicher M, Mueller MD, Hornung R, Fink D, Baessler K, Hampl M, Denhaerynck K, Spirig R, Engberg S. A patient-reported outcome measure to identify occurrence and distress of post-surgery symptoms of WOMen with vulvAr Neoplasia (WOMAN-PRO) - a cross sectional study. Gynecol Oncol. 2013 Apr;129(1):234-40. doi: 10.1016/j.ygyno.2012.12.038. Epub 2013 Jan 3. PMID 23290987
- [Background] Senn B, Mueller MD, Cignacco EL, Eicher M. Period prevalence and risk factors for postoperative short-term wound complications in vulvar cancer: a cross-sectional study. Int J Gynecol Cancer. 2010 May;20(4):646-54. doi: 10.1111/IGC.0b013e3181d92723. PMID 20686386
- [Background] Van der Zee AG, Oonk MH, De Hullu JA, Ansink AC, Vergote I, Verheijen RH, Maggioni A, Gaarenstroom KN, Baldwin PJ, Van Dorst EB, Van der Velden J, Hermans RH, van der Putten H, Drouin P, Schneider A, Sluiter WJ. Sentinel node dissection is safe in the treatment of early-stage vulvar cancer. J Clin Oncol. 2008 Feb 20;26(6):884-9. doi: 10.1200/JCO.2007.14.0566. PMID 18281661
- [Background] Senn, B., Gafner, D., Raphaelis, S., Meyer, G., Mayer, H., White, K.,. . . Mueller, M. D. (2013). Testing the counsellig program
- [Background] Lincoln, Y. S., & Guba, E. G. (1985). Naturalistic inquiry. Beverly Hills, Calif.: Sage Publications.
- [Background] Hampl, M., & Janni, W. (2012). Vulvakarzinom. Der Gynäkologe, 45(11), 865-872. https://doi.org/10.1007/s00129-012-2995-8
- [Background] Grove, S. K., Burns, N. P. D., & Gray, J. 1. (2012). The practice of nursing research: Appraisal, synthesis, and generation of evidence (7. ed.). Philadelphia Pa., London: Saunders.
- [Background] Flick, U. (2014). An introduction to qualitative research (Ed. 5). Los Angeles, Calif.: Sage.
- [Background] Dresing, T., & Pehl, T. (2011). Praxisbuch Transkription: Regelsysteme, Software und praktische Anleitungen für qualitative ForscherInnen (2. Auflage, Sept. 2011). Marburg: Eigenverlag.
- [Background] Denzin, N. K., & Lincoln, Y. S. (2011). The Sage handbook of qualitative research (4th ed.). Thousand Oaks: Sage.
- [Background] Creswell, J. W., & Plano Clark, V. L. (2017). Designing and conducting mixed methods research (3rd ed.). Los Angeles: Sage Publications.
- [Background] Anders, S., Riethdorf, L., & Löning, T. (2001). Neoplasia and pre-neoplasia of the lower genital tract. Der Gynäkologe, 34(7), 590-598. https://doi.org/10.1007/s001290101061
- See also: Royal College of Obstetricians and Gynaecologists. (2014). Guideline for Diagnosis and Management of Vulval Carcinoma. — https://www.rcog.org.uk/globalassets/documents/guidelines/vulvalcancerguideline.pdf
- See also: Swiss Confederation. (2014). Federal Law on Data Protection. — https://www.admin.ch/opc/de/classified-compilation/19920153/201401010000/235.1.pdf